CLINICAL TRIAL: NCT01688206
Title: An Open-label, Multi-center, Dose Escalation Phase I Study of Single Agent RO5520985 (Vanucizumab), and in Combination With Atezolizumab, Administered as an Intravenous Infusion in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of Vanucizumab (RO5520985) Alone or in Combination With Atezolizumab in Participants With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP28179; 2011-005877-22 (EudraCT Number); RG7221 (Other: Roche)
Record Dates: First submitted 2012-09-13; First posted 2012-09-19 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; vanucizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vanucizumab (Experimental): Participants will receive escalating doses of vanucizumab and fixed dose of vanucizumab, intravenously every 2 weeks.
  Interventions: Biological: Vanucizumab
- Vanucizumab + Atezolizumab (Experimental): Participants will receive fixed dose of vanucizumab along with atezolizumab, intravenously every 2 weeks.
  Interventions: Biological: Atezolizumab [TECENTRIQ]; Biological: Vanucizumab

INTERVENTIONS:
Biological: Atezolizumab [TECENTRIQ] — Participants will receive atezolizumab at a fixed dose of 840 mg, intravenously every 2 weeks.
  Other Names: RO5541267
  Arms: Vanucizumab + Atezolizumab
Biological: Vanucizumab — Participants will receive escalating doses of vanucizumab (starting dose: 3 milligram [mg] per kilogram) and fixed dose of vanucizumab (MTD/RP2D: 30 mg/kg), intravenously every 2 weeks.
  Other Names: RO5520985

SUMMARY:
This multi-center, open-label study will evaluate the safety, pharmacokinetics, pharmacodynamics and preliminary efficacy of vanucizumab as a single agent or in combination with atezolizumab in participants with locally advanced or metastatic solid tumors. Cohorts of participants will receive escalating doses of vanucizumab, fixed dose of vanucizumab (MTD and/or recommended phase two dose [RP2D]), and fixed dose of vanucizumab in combination with atezolizumab, intravenously every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed epithelial ovarian, fallopian tube or primary peritoneal cancer
* Participants must have platinum resistant disease defined as progression within <6 months from completion of a minimum of 4 platinum therapy cycles OR Participants must have platinum refractory disease, which is defined as progression during platinum based chemotherapy
* Less than or equal to (<=) 2 prior lines of systemic therapy
* The participant is willing to consent to and undergo a pre-treatment and on treatment core or excisional biopsy of the tumor
* Measurable disease as determined by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Adequate hematological function
* Adequate liver function
* Adequate renal function
* Adequate coagulation
* Adequate cardiovascular function
* Recovery from all reversible adverse events of previous anti-cancer therapies to baseline or Common Terminology Criteria for Adverse Events (CTCAE) Grade (G) 1, except for alopecia (any grade) and <= G 2 sensory peripheral neuropathy

Exclusion Criteria:

* Participants with primary central nervous system (CNS) tumors or CNS tumor involvement. Participants with metastatic CNS tumors may participate in this trial under conditions defined by protocol
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 of Cycle 1, or abdominal surgery, abdominal interventions or significant abdominal traumatic injury within 60 days prior to Day 1 of Cycle 1 or anticipation of the need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure
* Significant cardiovascular/cerebrovascular disease within 6 months prior to study drug administration
* Known human immuno deficiency virus (HIV) infection or known active hepatitis B or hepatitis C virus infection or active tuberculosis
* Participants previously treated with vascular endothelial growth factor (VEGF)-A inhibitors and with agents targeting Angiopoietin (Ang)-1/2 and/or Tyrosine-protein kinase receptor2
* History of intra-abdominal inflammatory process within the last 12 months such as, but not limited to, diverticulitis, peptic ulcer disease, or colitis
* Any prior radiotherapy to the pelvis or abdomen
* Treatment with systemic immunostimulatory agents, including but not limited to, interferon (IFN)-alpha, IFN-beta, interleukin (IL)-2, conjugated IL-2 cytokines within 6 weeks or five half-lives of the drug, whichever is longer, prior to screening
* History of bowel obstruction and/or clinical signs or symptoms of gastro-intestinal obstruction, including sub-occlusive disease related to the underlying disease (however, participants with signs/symptoms of sub/occlusive syndrome/bowel obstruction at the time of initial diagnosis may be enrolled if they had received definitive [surgical] treatment for symptom resolution). History of abdominal fistula or tracheo-oesophageal fistula, gastrointestinal perforation or intra-abdominal abscess, unless occurred and resolved before initial diagnosis and unrelated to the underlying cancer disease. Evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on Computed tomography (CT)
* Chronic daily treatment with non-steroidal anti-inflammatory drug (NSAID) (occasional use for the symptomatic relief of medical conditions, for example, headache, fever is allowed)
* Treatment with systemic immunosuppressive medications including, but not limited, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents within 2 weeks prior to study drug administration
* Previous treatment with checkpoint inhibitors (e.g. anti Programmed death [PD]-1, anti-PD-ligand 1, anti Cytotoxic T-lymphocyte-associated molecule-4) or prior treatment with cluster of differentiation (CD) 137 agonists or any other antibody or drug targeting T cell co-stimulation or other immune checkpoint blockade therapies
* History of autoimmune disease including, but not limited to systemic lupus erythematosus (SLE), Sjögren's syndrome, glomerulonephritis, multiple sclerosis, rheumatoid arthritis, vasculitis, systemic immune activation, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Guillain-Barré syndrome, Bell's palsy
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g. bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* Prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Administration of a live, attenuated vaccine within 4 weeks before Cycle1 Day1 or anticipation that such a live attenuated vaccine will be required during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Vanucizumab | approximately 28 days
Number of Participants With Objective Response According to RECIST 1.1 Criteria | approximately 3 years
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | approximately 3 years
Number of Participants With Dose-limiting Toxicities (DLTs) | approximately 28 days

SECONDARY OUTCOMES:
Elimination Half-life (t1/2) of Vanucizumab | Cycle 1 & 4: 0 hour (pre-dose), end of infusion (maximum up to 120 minutes); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)
Area Under the Plasma Concentration-time Curve During one Dosing Interval (AUCtau) of Vanucizumab | Cycle 1 & 4: 0 hour (pre-dose), end of infusion (maximum up to 120 minutes); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)
Clearance of Study Drug From the Body (CL) | Cycle 1 & 4: 0 hour (pre-dose), end of infusion (maximum up to 120 minutes); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)
Volume of Distribution at Steady-State (Vss) of Vanucizumab | Cycle 1 & 4: 0 hour (pre-dose), end of infusion (maximum up to 120 minutes); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)
Accumulation Ratio (RA) of Vanucizumab | Cycle 1 & 4: 0 hour (pre-dose), end of infusion (maximum up to 120 minutes); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)
Number of Participants With Objective Response According to RECIST 1.1 Criteria, CA-125 Response Criteria, and Immune-modified RECIST Criteria | approximately 3 years
Number of Participants With Disease Control According to RECIST 1.1 Criteria | approximately 3 years
Progression Free Survival (PFS) According to RECIST 1.1 Criteria | Baseline until disease progression or death (up to approximately 3 years)
Biological Progression-free Interval (PFIbio) According to RECIST 1.1 Criteria | Baseline until biologic progression or death (up to approximately 3 years)
Overall Survival (OS) | Baseline until death (up to approximately 3 years)
Change From Baseline in Micro Vessel Density (MVD) Assessed by Paired Tumor Biopsies | approximately 2 years
Change From Baseline in Proliferation and Apoptosis of Endothelial cells and Tumor Cells Assessed by Paired Tumor Biopsies | approximately 2 years
Change From Baseline in Maturity of Blood Vessels Assessed by Paired Tumor Biopsies | approximately 2 years
Change From Baseline in Targets and Receptors Assessed by Paired Tumor Biopsies | approximately 2 years
Change From Baseline in Blood Plasma Volume (Vp), Extracellular Extravascular Space Volume (Ve), and Volume Transfer Coefficient, Assessed by Bio-Imaging | approximately 2 years
Change From Baseline in Apparent Diffusion Coefficient (ADC) Assessed by Bio-Imaging | approximately 2 years
Percentage of Participants With Human Anti-Human Antibodies (HAHA) to Vanucizumab and Atezolizumab (ATA) | 0 hours (pre-dose) in Part I, II, and III (Cycle 1, 5, 6, end of study [EoS] visit) Part IV (Cycle 1, 3, 4, 8, every 8 weeks after cycle 8, EoS visit)
Area under the Concentration-time Curve (AUC) of Vanucizumab | Cycle 1 & 4: 0 hour (pre-dose), end of infusion (maximum up to 120 minutes); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)
Maximum Observed Plasma Concentration (Cmax) of Vanucizumab | Cycle 1 & 4: 0 hour (pre-dose), end of infusion (maximum up to 120 minutes); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)
Minimum Observed Plasma Concentration (Cmin) of Vanucizumab | Cycle 1 & 4: 0 hour (pre-dose); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)
Time of Observed Maximum Plasma Concentration (Tmax) | Cycle 1 & 4: 0 hour (pre-dose), end of infusion (maximum up to 120 minutes); Cycle 2, 3, 8, every 8 weeks after cycle 8: 0 hour (pre-dose)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Belgium (2):
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
- France (6):
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Francois Baclesse; Oncologie, Caen
  - Centre Leon Berard; Departement Oncologie Medicale, Lyon
  - Institut Curie; Oncologie Medicale, Paris
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut Gustave Roussy; Sitep, Villejuif
- Spain (6):
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia